CLINICAL TRIAL: NCT06539676
Title: A Prospective, Two-armed, Multicenter Clinical Study to Evaluate Efficacy, Performance, and Safety of Nighttime Aligners (Worn 10-12 Hours Day or Night) Compared to Daytime Aligners (Worn 20-22 Hours Day/Night)
Brief Title: A Study to Compare Nighttime Aligners to Daytime Aligners
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision to terminate study.
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-OR-24-017
Record Dates: First submitted 2024-06-28; First posted 2024-08-06 (Actual); Results first posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-06

CONDITIONS: Teeth Straightening; Aligner Therapy; Orthodontic Aligner

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nighttime Aligners (Experimental): Nighttime Aligners worn 10-12 hours per day or night
  Interventions: Device: Nighttime Aligners
- Daytime Aligners (Active Comparator): Daytime aligners worn 20-22 hours day and night
  Interventions: Device: Daytime Aligners

INTERVENTIONS:
Device: Nighttime Aligners — Nighttime aligners worn 10-12 hours per day or night during 2-8 months
  Arms: Nighttime Aligners
Device: Daytime Aligners — Daytime aligners worn 20-22 hours per day or night during 2-8 months
  Arms: Daytime Aligners

SUMMARY:
The purpose of this research study is to see if Nighttime Aligners (worn 10-12 hours per day or night) are effective and safe for tooth movement and if so, how they compare with the standard Daytime aligners (worn 20-22 hours per day), in adults and children from 12 years of age and older.

It will investigate the efficacy and performance of the treatments, as well as the safety of the investigational device and comparator.

The main objectives are:

* Comparison between the two groups concerning actual vs planned tooth movements (measured by changes in tooth position)
* Comparison between the two groups concerning the incidence of device or dental related AEs.
* Overall dentist and participant satisfaction with the treatment.

Participants will:

* Be given orthodontic aligner therapy with the Daytime (20-22h/day) or Nighttime (10-12h/day) Aligners (randomly assigned)
* Attend approximately 5 study during approximately 8-10 months

ELIGIBILITY:
Inclusion Criteria:

1. Subject willing to participate in the clinical study and able to understand the content of the clinical study.
2. Subject must have permanent dentition (i.e. all second molars).
3. Subject must be 12 years of age or older.
4. Subject must be able to provide and sign consent for themselves, without requiring consent to be given by a legally authorized representative. Parental consent is also required for all participants who are not of the legal age to provide consent themselves (based on participant state of residence).
5. The subject requires correction of teeth without planned extrusive movements on either or both arches.
6. The subject has no greater than 5 mm of crowding and/or spacing (based on estimation by Investigator).
7. The subject does not require planned correction of molar tooth positions, posterior bite or molar classic relationship corrections. Subjects with Class II or Class III malocclusions requiring posterior bite / class correction are not eligible.
8. Subjects without prior orthodontic treatment within the past 18 months.
9. Subjects who are periodontally stable.
10. Subjects without a known history of plastic allergies.
11. Subjects who have not had or do not require tooth extractions in preparation for orthodontic treatment with aligners.
12. Subjects with a treatment plan that does not include the use of elastics.

Exclusion Criteria:

1. Unlikely to be able to comply with clinical study procedures according to Investigator's judgement.
2. Unable or unwilling to return for follow-up visits.
3. Previous enrolment in the present clinical study.
4. Involvement in the planning and conduct of the clinical study (applies to both Sponsor personnel and the clinical study site)
5. Participation in another clinical study that may interfere with the present clinical study.
6. Subjects who have active carries, where there is no plan to correct them prior to the start of aligner therapy.
7. Other dental or clinical pathologies, which in the judgment of the Investigator, deem the candidates inappropriate for participation in the study (e.g. clinically significant periodontal disease or gingivitis, interproximal decay, etc.).
8. The subject require interproximal reduction or attachments to obtain a corrected malocclusion.
9. In addition to the criteria listed above, this product is contraindicated for use in adult and adolescent subjects presenting with the following dental conditions:

   * Active periodontal disease
   * Severe open bite or severe overjet
   * Tooth malocclusion requiring surgical correction
   * Subject with mixed dentition
   * Subject with a skeletally narrow jaw
   * Dental prosthetics/implants or significant number of missing teeth
10. Known pregnancy, pregnancy tests will be performed as per local requirements.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-01-17 (Actual); Study Completion 2025-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay Khorsandi, Dr, Study Director — BYTE
Locations (12):
- United States (12):
  - Fulbright Dental, Redondo Beach, California
  - 3D Dental, Miami Beach, Florida
  - Elite Dental of Towson, Towson, Maryland
  - Cedars Family Dental, Plainville, Massachusetts
  - R. Lobato & Associates, Las Vegas, Nevada
  - Aesthetic Dental, North Bergen, New Jersey
  - Huerta Dentistry, New York, New York
  - Brush365, Frisco, Texas
  - Gustafson Dental, Humble, Texas
  - SKM Dentistry d/b/a brush365 Dental, Hurst, Texas
  - Northwest Dental Medicine, Puyallup, Washington
  - Gregson Family Dentistry, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study was terminated early. At time of study termination seven (7) subjects had been consented (started), out of which only one subject had been randomised and allocated a treatment arm (Treatment Start Visit). To report the six (6) subjects not yet assigned a treatment arm at time of early study termination, an additional Arm "Treatment Not assigned" was included.
Groups:
- Treatment Not Assigned: Subjects consented but where no treatment was assigned prior to early study termination.
Period: Overall Study
Arm/Group | Nighttime Aligners | Daytime Aligners | Treatment Not Assigned
Started | 1 | 0 | 6
Treatment Start Visit | 1 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 1 | 0 | 6
Not completed — Early study termination | 1 | 0 | 6

BASELINE CHARACTERISTICS:
Population: All screened subjects.
  This study was terminated early. At time of study termination seven (7) subjects had been consented, out of which only one subject had been randomised and allocated a treatment arm. To present Results Baseline Characteristics for all screened subjects, the two planned treatment arms have been combined into one.
Groups:
- Aligners: Either Nighttime Aligners worn 10-12 hours per day or night, or daytime aligners worn 20-22 hours day and night
Arm/Group | Aligners
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: Years] | 32.4 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Peer Assessment Rating (PAR) Index
Description: Comparison between actual vs planned tooth movements, compared between the investigational treatment and the control device
Time Frame: From day 0 (Treatment start) up to 8 months post treatment start (Final visit)
Population: No subject conducted the final visit prior to early study termination. Consequently, no outcome data has been obtained in the study for this outcome and can thus not be presented.
Arm/Group | Nighttime Aligners | Daytime Aligners
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Subject Satisfaction With the Treatment
Description: Overall subject satisfaction with the treatment assessed by a questionnaire using a rating scale from 1 to 10 (1 very satisfied - 10 very unsatisfied).
Time Frame: At the final visit (2-8 months post day 0)
Population: as for outcome 1
Arm/Group | Nighttime Aligners | Daytime Aligners
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Dentist (Investigator) Satisfaction With the Treatment
Description: Overall dentist (investigator) satisfaction with the treatment assessed by a questionnaire using a rating scale from 1 to 10 (1 very satisfied - 10 very unsatisfied).
Time Frame: At the final visit (2-8 months post day 0)
Population: as for outcome 1
Arm/Group | Nighttime Aligners | Daytime Aligners
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Subject Self-reported Pain/Discomfort
Description: The subject self-reported values pertaining to pain/discomfort during treatment and comfort in wearing the aligners captured in a questionnaire with Visual Analogue Scale (VAS) with a Wong Baker face scale (score 0-10), where a higher score corresponds to a higher level of pain/discomfort.
Time Frame: At each follow-up visit (Follow-up visits every 4-6 weeks post Day 0 during a 2-8 months period) and at the final visit (Day 0 + 2-8 months).
Population: All subjects allocated a treatment arm (one subject in total).
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Nighttime Aligners | Daytime Aligners
Number analyzed (Participants) | 1 | 0
score on a scale
  Visit 1. Between this visit and the previous visit, how comfortable are the aligners to wear | 9 [9 to 9] |
  Visit 2. Between this visit and the previous visit, how comfortable are the aligners to wear | 9 [9 to 9] |
  Visit 3. Between this visit and the previous visit, how comfortable are the aligners to wear | 0 [0 to 0] |
  Visit 1. Pain associated with new tooth movement between this visit and the previous visit | 0 [0 to 0] |
  Visit 2. Pain associated with new tooth movement between this visit and the previous visit | 0 [0 to 0] |
  Visit 3. Pain associated with new tooth movement between this visit and the previous visit | 0 [0 to 0] |

ADVERSE EVENTS:
Time Frame: From informed consent up to study termination (up to 4.5 months).
Description: This study was terminated early. At time of study termination seven (7) subjects had been consented (started), out of which only one subject had been randomised and allocated a treatment arm (Treatment Start Visit). To report the six (6) subjects not yet assigned a treatment arm, an additional Arm "Treatment Not assigned" was included.
Arm/Group | Nighttime Aligners | Daytime Aligners | Treatment Not Assigned
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/6
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nighttime Aligners (N=1) | Daytime Aligners (N=0) | Treatment Not Assigned (N=6)
Chipped bonding on a front tooth (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — Patient chipped bonding on a front tooth when she was eating a candy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/76/NCT06539676/Prot_SAP_001.pdf